CLINICAL TRIAL: NCT00426348
Title: A Prospective Randomized, Controlled, Double Blinded Trial of the Antioxidant Probucol Combined With Valsartan in Patients With IgA Nephropathy
Brief Title: A Study of the Antioxidant Probucol Combined With Valsartan in Patients With IgA Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Shi, Director of renal division of Guangdong General Hospital, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPPH200603
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Glomerulonephritis; IGA Nephropathy
Keywords: IgA nephropathy; probucol; valsartan; treatment; antioxidant; IGA nephropathy：a kind of glomerulonephritis,which IgA is the dominant immunodeposit in mesangial areas
MeSH Terms: conditions — Glomerulonephritis; Glomerulonephritis, IGA | interventions — Valsartan; Probucol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): In arm 1,Valsartan(80-160mg/day) is given to patients in combination with Placebo
  Interventions: Drug: Valsartan; Drug: Placebo
- 2 (Experimental): Valsartan(80-160mg/day) + Probucol(750mg/day)
  Interventions: Drug: Valsartan; Drug: Probucol

INTERVENTIONS:
Drug: Valsartan — Valsartan (80-160mg/day)
Drug: Probucol — Probucol (750mg/day)
  Arms: 2
Drug: Placebo — Placebo
  Arms: 1

SUMMARY:
a statement of the study hypothesis:the effect of valsartan in patients with IgA nephropathy have been proved,and the efficacy of probucol in combination with valsartan is to be proved in patients with IgA nephropathy.

This is a prospective randomized controlled, double blinded pilot study to identify the efficacy of probucol in combination with valsartan in patients with IgA nephropathy. The renal function deterioration will be the primary outcome studied. The expected study duration will be 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill the clinical and pathological criteria for IgA nephropathy
* Age: 18-60 years
* Renal biopsy diagnostic for IgA nephropathy based on immunohistologic staining for IgA that is greater than or equal to staining for IgG and IgM
* Urinary protein excretion rate is within the range of 1-2.5g/day
* Serum creatinine <265.2umol/L at the time of randomization

Exclusion Criteria:

* Patients who refuse to be randomized for treatment
* Patients who prefer treatment with conventional agents
* Patients who are pregnant or plan for pregnancy
* Patients who are pathologically proven severely or diffusely proliferative IgA nephropathy or crescent glomerulonephritis with >= 50% segmental involvement of the glomeruli and should be treated with other agents,such as immunosuppressive agents or steroid
* Clinical and histologic evidence of:

  * systemic lupus erythematosus
  * Henoch-Schonlein purpura
  * cirrhosis
  * chronic active liver disease
  * hepatitis B
  * hepatitis C
  * severe chronic diarrhea
  * active peptic ulcer disease
  * HIV
  * acute renal failure
  * malignant hypertension
  * severe heart diseases
  * malignant tumor
  * any systemic infection
  * pregnancy
  * Known contraindication to the administration of probucol and valsartan

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2007-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
urinary protein loss whithin 24 hours | 2-3years

SECONDARY OUTCOMES:
renal function(serum Crea or eGFR) deterioration | 2-3years

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, PhD,MD, Principal Investigator — Nephrology Dept.,Guangdong General Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Ye Z, Zhang L, Xu L, Shi W, Hu H, Shi X, Zhong W, Hou S, Yan H, Zhang B, Xia Y, Wang W, Feng Z, Wang L, Liang Y. Probucol combined with valsartan in immunoglobulin A nephropathy: a multi-centre, open labelled, randomized controlled study. Nephrology (Carlton). 2014 Jan;19(1):40-6. doi: 10.1111/nep.12177. PMID 24191893